CLINICAL TRIAL: NCT02099864
Title: Molecular Mechanisms Underlying Tumor Progression Despite Enzalutamide Treatment
Brief Title: Genetic and Molecular Mechanisms in Assessing Response in Patients With Prostate Cancer Receiving Enzalutamide Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Astellas Pharma US, Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alexandra Sokolova, M.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00010241; NCI-2014-00417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IIT000800; MR00045569; IRB00010241 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Soft Tissues; Metastatic Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage III Prostate Adenocarcinoma AJCC v7; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Enzalutamide) (Experimental): Patients receive enzalutamide PO QD in the absence of disease progression or unacceptable toxicity. Patients undergo a tumor biopsy of a metastatic site at study entry (prior to initiation of enzalutamide) and after the time of progression. Per the investigator, patients may continue treatment beyond progression.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi

SUMMARY:
This phase II trial studies genetic and molecular mechanisms in assessing response in patients with prostate cancer receiving enzalutamide therapy. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as enzalutamide, may lessen the amount of androgens made by the body. Studying samples of tissue and blood in the laboratory from patients with prostate cancer may help doctors better understand castration-resistant prostate cancer. It may also help doctors make improvements in prostate cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the correlations between baseline molecular features and pathways and prostate-specific antigen (PSA) change (</>= 50% decline) at 12 weeks versus (vs.) baseline.

SECONDARY OBJECTIVES:

I. To measure PSA change at 12 weeks and at each study visit vs. baseline after enzalutamide treatment.

II. To measure objective response after enzalutamide treatment. III. To assess the correlations between the baseline molecular features and pathways and progression-free survival, disease-specific survival, and overall survival.

IV. To assess the correlations between the baseline molecular features and pathways and time to PSA progression.

V. To identify molecular features and cellular pathways present in tumors from men with metastatic castrate-resistant prostate cancer (CRPC) that are progressing despite enzalutamide treatment.

VI. To explore correlation between baseline molecular features and pathways and changes in circulating tumor cells (CTCs) counts.

VII. To explore correlation between baseline molecular features and pathways and objective response.

VIII. To assess the correlations between the baseline molecular features and pathways and degree of PSA decline at 12 weeks and maximal PSA decline observed while on study.

IX. To assess the correlations between the baseline molecular features and time on treatment.

EXPLORATORY OBJECTIVES:

I. To assess correlations between cell-free deoxyribonucleic acid (DNA) (cfDNA) molecular features from blood and molecular features and pathways from the biopsy samples.

II. To assess correlations between cfDNA molecular features and endpoints in the primary and secondary objectives listed above.

III. To assess correlations between cell-free DNA and tumor molecular features and changes in PSA after discontinuing enzalutamide.

IV. To explore correlations with baseline molecular features and tissue histology.

V. To explore correlations with baseline tissue histology and PSA change, time to PSA progression, time on treatment, progression-free survival, and overall survival.

OUTLINE:

Patients receive enzalutamide orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity. Patients undergo a tumor biopsy of a metastatic site at study entry (prior to initiation of enzalutamide) and after the time of progression. Patients may continue treatment beyond progression at the investigator's discretion.

After completion of study treatment, patients are followed up at 2-3 or 6 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without pure small cell carcinoma; patients without histologically confirmed adenocarcinoma may be eligible if both the treating physician and the study principal investigator (PI) agree that the patient's history is unambiguously indicative of advanced adenocarcinoma
* Ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration); patients who have not had an orchiectomy must maintain effective GnRH-analogue therapy for the duration of the trial
* Radiographic evidence of regional or distant metastases with suspected tumor in an area that is safe to biopsy
* Willingness to undergo a tumor biopsy at baseline and at disease progression
* Serum testosterone level < 50 ng/dL at screening
* Progressive disease by PSA or imaging in the setting of medical or surgical castration; disease progression for study entry is defined as one or more of the following three criteria:

  * PSA evidence for progressive prostate cancer which consists of a PSA level of at least 2 ng/ml which has risen on at least 2 successive occasions, at least 1 week apart; if the confirmatory PSA value is less than the screening value, then an additional PSA value greater than #2 will be required to document progression of >= 1 week

    * PSA values to be obtained >= 1 week apart
  * Soft tissue disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
  * Bone disease progression defined by two or more new lesions on bone scan
* Patient's physician has already recommended enzalutamide for treatment of progression
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Willing and able to give informed consent
* Estimated life expectancy >= 6 months
* Subjects who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last study drug administration
* A minimum of 4 weeks elapsed off of anti-androgen therapy prior to enrollment for flutamide and 6 weeks for bicalutamide and nilutamide without evidence of an anti-androgen withdrawal response; patients who NEVER HAD A PSA decline with the most recent anti-androgen therapy or in whom the response to the most recent anti-androgen was for < 3 months require only a 2 week washout period prior to first dose of study drug
* A minimum of 4 weeks from prior systemic anti-cancer therapies or 3 weeks for radiation treatment prior to enrollment is required

Exclusion Criteria:

* Severe, concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment
* Previous treatment with docetaxel for metastatic prostate cancer
* Known metastases in the brain or active epidural disease (NOTE: patients with treated epidural disease are allowed)
* Absolute neutrophil count < 1,000/uL
* Platelet count < 75,000/uL
* Hemoglobin < 9 g/dL at the screening visit; (NOTE: subject may not have received any growth factors or blood transfusions within seven days of the hematologic laboratory values obtained at the screening visit)
* Total bilirubin (TBL) > 2.5 times the upper limit of normal at the screening visit
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal at the screening visit
* Creatinine (Cr) > 2 mg/dL at the screening visit
* Prothrombin time (PT) or international normalized ratio (INR) and a partial thromboplastin time (PTT) > 1.5 times the upper limit of normal
* Previous treatment with an agent that blocks adrenal androgen synthesis (e.g. abiraterone acetate, TAK-700, TOK-001, ketoconazole) or second generation androgen receptor (AR) antagonists (e.g., BMS 641988, ARN-509,TOK-001)
* Systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within 4 weeks of study drug administration are prohibited
* Structurally unstable bone lesions suggesting impending fracture
* Previous treatment with enzalutamide (MDV3100)
* Medical contraindications to stopping aspirin, Coumadin or other anticoagulants prior to image-guided tumor biopsies; follow institutional guidelines when determining drugs to avoid and length of washout
* Plans to initiate treatment with an investigational agent during the study
* History of seizure or condition that may predispose to seizure; also, history of loss of consciousness or transient ischemic attack within 12 months of (day 1 visit)
* Concomitant use of the strong CYP2C8 inhibitors gemfibrozil or trimethoprim (Bactrim)
* History of known malabsorption syndrome or prior surgery(ies) that may lead to malabsorption
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) within 4 weeks of study drug administration (day 1)
* Use of the following drugs within 4 weeks of study drug administration: 5 alpha-reductase inhibitors (finasteride, dutasteride), estrogens, Cyproterone acetate, biologic, or other agents with anti-tumor activity against prostate cancer, and androgens (testosterone, dihydroepiandrosterone [DHEA], etc.)
* A second active malignancy except adequately treated non-melanoma skin cancer or other non-invasive or in situ neoplasm

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sokolova, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - OHSU Knight Cancer Institute, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzalutamide)
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 29
Age, Continuous [Median (Full Range); unit: years] | 71.9 [56.6 to 88.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a >= 50% Decline in Prostate-specific Antigen (PSA) Value
Description: The percentage of participants with a >= 50% decline in PSA values will be reported with 95% exact confidence interval. For each participant, percentage decline in PSA values are calculated as 100% times the difference between PSA values taken at baseline and 12 weeks divided by PSA values at baseline. Percentage of participants determined as 100% times the number of participants with >= 50% decline divided by overall number of participants.
Time Frame: Baseline to 12 weeks
Population: Evaluable patients will include those patients for whom data from genomic studies and IHC tests are available from the pre-treatment biopsy samples and who have completed at least 12 weeks of therapy or who have confirmed disease progression prior to 12 weeks of therapy, and for whom baseline and 12 week PSA data were available. 36 subjects shown in participant flow. 2 subjects were excluded from this PSA analysis: 1 had missing PSA data, 1 had falling PSA in setting of rapid disease progression
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 34
percentage of subjects | 73.5 [55.6 to 87.1]

2. Primary Outcome: Percentage of Participants With Tumor Protein 53 Gene (TP53) Copy Number Alterations and Mutations
Description: Evaluate the association between PSA response at 12 weeks after initiating therapy, and TP53 copy number alterations and mutations at baseline. Simple Logistic regression was planned but due to sample size we used Fisher's Exact test. Percentage of patients in each arm with TP53 copy number alterations and mutations will be reported and odds ratio with two-sided 95% confidence interval will be calculated.
Time Frame: Baseline to 12 weeks
Population: For the primary endpoint, evaluable patients will include those patients for whom data from genomic studies and IHC tests are available from the pre-treatment biopsy samples and who have completed at least 12 weeks of therapy or who have confirmed disease progression prior to 12 weeks of therapy. Targeted DNA sequencing was performed on 26 of 36 biopsies that contained sufficient material.
Measure: Number; unit: percentage of subjects
Groups:
- Responders: PSA Responder: A ≥ 50% reduction at 12 weeks after the initiation of therapy vs. baseline. Baseline PSA will be defined as the measurement obtained immediately prior to initiation of Enzalutamide on Day 1 of study.
- PSA Non-responders: PSA Non-Responder: A less than 50% reduction at 12 weeks after the initiation of therapy vs. baseline. Baseline PSA will be defined as the measurement obtained immediately prior to initiation of Enzalutamide on Day 1 of study.
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 21 | 5
percentage of subjects | 28.6 | 80.0
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p = 0.055, Fisher Exact; Due to sample size, Fisher's exact test was used rather than simple logistic regression; Odds Ratio (OR) = 10.0, 95% CI 2-sided [0.9 to 108.8]

3. Primary Outcome: Percentage of Participants With Phosphatase and Tensin Homologue Gene (PTEN) Copy Number Alterations and Mutations
Description: Evaluate the association between PSA response at 12 weeks after initiating therapy, and PTEN copy number alterations and mutations at baseline. Simple Logistic regression was planned but due to sample size we used Fisher's Exact test. Percentage of patients in each arm with PTEN copy number alterations and mutations will be reported and odds ratio with two-sided 95% confidence interval will be calculated.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 21 | 5
percentage of subjects | 47.6 | 40.0
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p = 1.000, Fisher Exact; Due to sample size, Fisher's exact was used rather than regression; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.1 to 5.3]

4. Primary Outcome: Percentage of Participants With Retinoblastoma Gene (RB1) Copy Number Alterations and Mutations
Description: Evaluate the association between PSA response at 12 weeks after initiating therapy, and RB1 copy number alterations and mutations at baseline. Simple Logistic regression was planned but due to sample size we used Fisher's Exact test. Percentage of patients in each arm with RB1 copy number alterations and mutations will be reported and odds ratio with two-sided 95% confidence interval will be calculated.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 21 | 5
percentage of subjects | 9.5 | 0.0
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.0 to 17.0]

5. Primary Outcome: Androgen Receptor (AR) Messenger RNA (mRNA) Expression
Description: Median AR mRNA expression between responders and non-responders.
Time Frame: Baseline to 12 weeks
Population: Evaluable patients will include those patients for whom data from genomic studies and IHC tests are available from the pre-treatment biopsy samples and who have completed at least 12 weeks of therapy or who have confirmed disease progression prior to 12 weeks of therapy, and for whom baseline and 12 week PSA data were available. RNA sequencing was performed on 25 of 36 biopsies that contained sufficient material.
Measure: Median (Standard Deviation); unit: TPM
Groups:
- Non-responders: PSA Non-Responder: A less than 50% reduction at 12 weeks after the initiation of therapy vs. baseline. Baseline PSA will be defined as the measurement obtained immediately prior to initiation of Enzalutamide on Day 1 of study.
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 18 | 7
TPM | 224.9 (133.2) | 201.7 (201.7)
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Other; p = 0.84, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 23.2 — Difference is the median for responders minus the median for non-responders

6. Primary Outcome: Androgen Receptor Variant 7 (AR-V7) Expression
Description: Median AR-V7 expression between responders and non-responders.
Time Frame: Baseline to 12 weeks
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: TPM
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 18 | 7
TPM | 10.4 (7.2) | 12.3 (11.8)
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.9 — Difference is the median for responders minus the median for non-responders

7. Primary Outcome: Percentage of Participants With Androgen Receptor (AR) Copy Number Alterations and Mutations
Description: Evaluate the association between PSA response at 12 weeks after initiating therapy, and AR copy number alterations and mutations at baseline. Simple Logistic regression was planned but due to sample size we used Fisher's Exact test. Percentage of patients in each arm with AR copy number alterations and mutations will be reported and odds ratio with two-sided 95% confidence interval will be calculated.
Time Frame: Baseline to 12 weeks
Population: For the primary endpoint, evaluable patients will include those patients for whom data from genomic studies and IHC tests are available from the pre-treatment biopsy samples and who have completed at least 12 weeks of therapy or who have confirmed disease progression prior to 12 weeks of therapy. AR immunohistochemistry was available in 22 patients with sufficient samples.
Measure: Number; unit: percentage of subjects
Groups:
- PSA Non-responders: PSA non-responders: A less than 50% reduction at 12 weeks after the initiation of therapy vs. baseline. Baseline PSA will be defined as the measurement obtained immediately prior to initiation of Enzalutamide on Day 1 of study.
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 19 | 3
percentage of subjects | 73.7 | 100.0
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p = 1.00, Fisher Exact; Odds Ratio (OR) = 2.7, 95% CI 2-sided [0.1 to 60.2]

8. Primary Outcome: Number of Participants With Protein Expression of AR
Description: The number of participants, responders and non-responders, that were found to have protein expression of AR.
Time Frame: Baseline to 12 weeks
Population: For the primary endpoint, evaluable patients will include those patients for whom data from genomic studies and IHC tests are available from the pre-treatment biopsy samples and who have completed at least 12 weeks of therapy or who have confirmed disease progression prior to 12 weeks of therapy. AR protein expression was analyzed using immunohistochemical analysis from 21 patients with sufficient samples.
Measure: Number; unit: participants
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 15 | 6
participants | 15 | 6

9. Primary Outcome: Androgen Receptor (AR) Activity Level
Description: Median Normalized Enrichment Score (NES) AR activity levels of responders and non-responders. Gene Set Enrichment Analysis (GSEA) is used to interpret gene expression data. GSEA enrichment score (ES) reflects the degree to which a gene set (GS) is overrepresented at the top or bottom of a ranked list of genes. ES is calculated by walking down the list, increasing a running-sum statistic when a gene is in the GS and decreasing when it's not. Magnitude of increment depends on correlation of the gene with the phenotype. ES is the max deviation from zero encountered in walking the list. Positive ES indicates GS enrichment at the top of the list; negative indicates GS enrichment at the bottom. GSEA calculates NES as actual ES divided by mean (ESs against all permutations of the dataset). Low AR activity has been linked to stemness and lineage plasticity that are recognized as a cause of acquired resistance to AR-targeting therapies.
Time Frame: Baseline to 12 weeks
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 18 | 7
score on a scale | 2.2 (3.3) | -2.6 (1.4)
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 4.8 — Difference is the median for the responders minus the median for the non-responders

10. Secondary Outcome: Prostate-specific Antigen (PSA) Changes
Description: Number of patients who achieved a 50% or greater PSA decline any time after 12 weeks post-baseline.
Time Frame: Baseline to up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 34
Participants | 25

11. Secondary Outcome: Percentage of Participants With an Objective Response
Description: The percentage of participants with an objective response will be reported with 95% exact confidence interval. Objective radiographic response is evaluated using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. For each participant, objective response is calculated as 100% times the difference between the sum of measurable target lesions at baseline and the smallest sum of measurable target lesions achieved after the initiation of therapy, divided by the sum of target lesions at baseline.
Time Frame: Baseline to date of first documented radiographic objective response, assessed up to 1 year
Population: Only those subjects who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for objective response.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Treatment (Enzalutamide)
Number analyzed (Participants) | 22
percentage of subjects | 63.6 [40.7 to 82.8]

12. Secondary Outcome: Progression-free Survival (PFS)
Description: Correlations between baseline molecular features and pathways and PFS will be assessed using cox regression model. In addition, Kaplan-Meier plots will be used to graphically illustrate the survival distributions across the strata of categorical molecular predictors.
Time Frame: Time from day 1 of study drug treatment to date of first documented radiographic progression or clinical progression, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 25 | 9
months | 23.9 [10.9 to 33.6] | 3.7 [2.0 to 11.0]
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.18, 95% CI 2-sided [0.07 to 0.45]

13. Secondary Outcome: Disease-specific Survival (DSS)
Description: Correlations between baseline molecular features and pathways and DSS will be assessed using cox regression model. In addition, Kaplan-Meier plots will be used to graphically illustrate the survival distributions across the strata of categorical molecular predictors.
Time Frame: Time from day 1 of study drug treatment to date of death from prostate cancer, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 29 | 9
months | 38.6 [21.3 to 45.1] | 16.0 [4.7 to 23.8]
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.08 to 0.56]

14. Secondary Outcome: Overall Survival (OS)
Description: Correlations between baseline molecular features and pathways and OS will be assessed using cox regression model. In addition, Kaplan-Meier plots will be used to graphically illustrate the survival distributions across the strata of categorical molecular predictors.
Time Frame: Time from day 1 of study drug treatment to date of death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 25 | 9
months | 36.90 [21.29 to NA] — Upper limit of confidence interval not estimable; there are not enough events at later times to get a reliable estimate. | 15.97 [4.65 to 23.80]
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p = 0.23, Regression, Cox; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.02 to 0.59]

15. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Correlations between baseline molecular features and pathways and time to PSA progression will be assessed.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 24 | 9
months | 23.9 [10.9 to 33.6] | 3.7 [2.0 to 11.0]
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.18, 95% CI 2-sided [0.07 to 0.45]

16. Secondary Outcome: Molecular Features and Cellular Pathways Present in Tumors That Are Progressing Despite Treatment With Enzalutamide
Description: Random Forests classification will be used to identify molecular features and pathways present in patients with disease progression or who discontinue Enzalutamide treatment.
Time Frame: Up to 5 years
Population: We did not perform a random forest classifier. Rather, we used gene set enrichment analysis to understand transcriptional differences between responders and non-responders.
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Changes in Circulating Tumor Cell (CTC) Counts
Description: Linear regression model will be used to assess the association for changes in CTC counts from baseline and maximal prostate-specific antigen (PSA) observed while on study.
Time Frame: Baseline to up to 5 years
Population: Data were not collected
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Degree of Prostate-specific Antigen (PSA) Decline
Description: Degree of prostate-specific antigen (PSA) change from baseline to 12 weeks. PSA at week 12 minus PSA at baseline divided by PSA at baseline and multiplied by 100%. Decline shown as negative percent and incline shown as positive percent.
Time Frame: At 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PSA at baseline
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 25 | 9
percentage of PSA at baseline | -86.7 (13.5) | 101.8 (140.2)

19. Secondary Outcome: Maximal Prostate-specific Antigen (PSA) Decline Observed
Description: Correlations between baseline molecular features and pathways and maximal PSA decline observed will be assessed. Linear regression model will be used to assess the association for changes in circulating tumor cells (CTC) counts from baseline and maximal PSA observed while on study.
Time Frame: Up to 5 years
Population: Data were not collected
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Time on Treatment
Description: The association between molecular predictors and survival outcomes (e.g., progression-free survival [PFS], disease-free survival [DSS] and overall survival [OS]) and time on treatment will be assessed using cox regression model.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Responders | PSA Non-responders
Number analyzed (Participants) | 25 | 9
months | 24.23 [11.55 to 40.35] | 3.43 [2.29 to 14.59]
Statistical Analysis 1: Comparison: Responders vs PSA Non-responders; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 4.90, 95% CI 2-sided [2.03 to 11.82]

ADVERSE EVENTS:
Time Frame: Median time period for adverse events 14 months (range 2 months to 53 months). Deaths assessed up to 5 years.
Description: Collected from the start date of treatment with enzalutamide to the last date of treatment with enzalutamide. Adverse events are collected for any untoward clinical experience with the exception of lab abnormalities which are only reported if the test result is deemed Clinically Significant by the responsible or treating physician. Clinical significance is based on clinical judgement and individual patient situation, at the discretion of the physician. Deaths assessed up to 5 years.
Arm/Group | Treatment (Enzalutamide)
All-Cause Mortality (participants affected / at risk) | 2/36
Serious Adverse Events (participants affected / at risk) | 6/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzalutamide) (N=36)
fracture (Injury, poisoning and procedural complications) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disease progression (General disorders) | 1
Heart failure (Cardiac disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Renal and urinary disorders - other, kidney cancer (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzalutamide) (N=36)
depression (Psychiatric disorders) | 3
diarrhea (Gastrointestinal disorders) | 3
dizziness (Nervous system disorders) | 4
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Dysgeusia (Nervous system disorders) | 3
edema limbs (General disorders) | 4
fall (Injury, poisoning and procedural complications) | 12
fracture (Injury, poisoning and procedural complications) | 9
Gynecomastia (Reproductive system and breast disorders) | 3
Hematuria (Renal and urinary disorders) | 3
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Nervous system disorders - Other, neuropathy (Nervous system disorders) | 3
pain (General disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
back pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, hip pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal and connective tissue disorder - Other, shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Paresthesia (Nervous system disorders) | 3
Presyncope (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 2
Stroke (Nervous system disorders) | 4
Upper respiratory infection (Infections and infestations) | 5
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 4
Weight loss (Investigations) | 2
fatigue (General disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02099864/Prot_SAP_000.pdf